CLINICAL TRIAL: NCT04548843
Title: A First in Human Phase I, Open Label Dose-escalation Study to Evaluate the Safety of Infusion of MNV-BM-PLC (Autologous CD34+ Cells Enriched With Placenta Derived Allogeneic Mitochondria) in Patients With Primary Mitochondrial Diseases Associated With Mitochondrial DNA Mutation or Deletion
Brief Title: A First in Human Study to Evaluate the Safety of Infusion of MNV-BM-PLC (Autologous CD34+ Cells Enriched With Placenta Derived Allogeneic Mitochondria) in Patients With Primary Mitochondrial Diseases Associated With Mitochondrial DNA Mutation or Deletion
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No recruitment
Sponsor: Minovia Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLC-PMD-01-IL
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Primary Mitochondrial Diseases
Keywords: Mitochondrial DNA Mutation or Deletion
MeSH Terms: interventions — Blood Component Removal

STUDY DESIGN:
Intervention Model Description: The study will involve two sequential cohorts:
  Cohort 1: 3 patients will be administrated with Dose 1 The dosing interval between patients will be at minimum 2 weeks. Two (2) weeks after the 3rd patient has received MNV-BM-PLC, the Data safety monitoring board (DSMB) will convene to review accumulated safety data. The DSMB will make a recommendation whether to proceed with the 4th patient administration.
  Cohort 2: 3 patients will be administrated with Dose 2 The dosing interval between patients will be at minimum 2 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 & Cohort 2 (Experimental): 3 patients will be administrated with Dose 1 (0.88 mitochondria unit (mU) citrate synthase (CS) activity per million cells).
  3 patients will be administrated with Dose 2 (4.4mU mitochondria unit (mU) citrate synthase (CS) activity per million cells).
  Interventions: Procedure: Bone Marrow mobilization; Procedure: Apheresis; Biological: MNV-BM-PLC infusion

INTERVENTIONS:
Procedure: Bone Marrow mobilization — During four days before the apheresis, Neupogen (G-CSF) at a dose of 10 microgram per kilogram will be administered subcutaneously in the morning (days -6 to -3 of cell therapy). In addition, Mozobil (Plerixafor) at a dose of 0.24 milligram per kilogram will be administered subcutaneously approximately 4 hours before apheresis initiation.
  A fifth dose of Neupogen (G-CSF) will be administered just prior to the apheresis
Procedure: Apheresis — Apheresis will be performed two days prior to MNV-BM-PLC infusion. During this procedure, patient's peripheral blood will be collected by apheresis
Biological: MNV-BM-PLC infusion — The MNV-BM-PLC (autologous CD34+ cells enriched with placenta-derived allogeneic mitochondria) infusion will be performed by standard IV procedure.
  The dosing interval between patients will be at minimum 2 weeks.

SUMMARY:
The study objectives are to evaluate the safety of a single intravenous (IV) infusion of autologous CD34+ cells enriched with placenta-derived allogeneic mitochondria in participant with primary mitochondrial disease associated with mitochondrial DNA mutations or deletions.

6 participants aged from 4 to 18 years old on the day of screening visit with primary mitochondrial disease associated with mitochondrial DNA mutations or deletions will be enrolled.

DETAILED DESCRIPTION:
MNV-BM-PLC is a personalized cell therapy based on autologous patient-derived Hematopoietic stem/progenitor cells (HSPCs) enriched with mitochondria isolated from healthy placenta obtained from donors during C-section. Healthy mitochondria are employed, ex-vivo, to enrich the patient's CD34+ peripheral blood cells, followed by infusion of the mitochondrial enriched cells back to the patient. This therapeutic process of mitochondrial augmentation provides the patient with healthy mitochondria carrying non-mutated/deleted mtDNA that can supplement mitochondrial functionality in the patient's cells.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of primary mitochondrial disease
* Age between 4 years and up to 18 years, with a minimum body weight of 20 (+/-1) kilogram on the day of screening visit.
* Performance score: Karnofsky ≥40 (or equivalent in children younger than 16 years old.
* Patients or Patient's parents or legal guardian (where applicable) has a good understanding of the study and nature of the procedure and is willing and able to provide written informed consent prior to participation in any study-related procedures.
* Medical ability to undergo the study procedures safely, as determined by the investigator.

Exclusion Criteria

* Positive test for pathogenic agents .
* Inability to undergo leukapheresis, as determined by the investigator.
* Chronic severe infection or any other disease or condition that may risk the patient or interfere with the ability to interpret the study results.
* Known history of malignancy.
* Patient has been treated within the last one year prior to IP treatment with a different cell therapy.
* Patient has participated in another interventional clinical study and/or received other experimental medication outside of a clinical study within 1 month prior the day of Investigation product (IP) treatment visit.
* A pregnant or lactating woman or a woman who plans to become pregnant during the study. In addition, any woman of childbearing potential (not sterile or postmenopausal), who is unwilling to adhere to the use highly effective contraception method for the duration of the study
* In the opinion of the Investigator, the patient is unsuitable for participating in the study due to safety concerns.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-related adverse events as assessed by CTCAE v5.0 following MNV-BM-PLC | 1 month
  Severity will graded according to CTCAE, Version 5.0
Measurement of hemoglobin level | 1 month
  Change from baseline in hematological parameter
Measurement of absolute neutrophil count | 1 month
  Change from baseline in hematological parameter
Measurement of platelet count | 1 month
  Change from baseline in hematological parameter

SECONDARY OUTCOMES:
Number of participants with Treatment-related adverse events as assessed by CTCAE v5.0 following MNV-BM-PLC | 2 years
  Severity will graded according to CTCAE, Version 5.0
Measurement of hemoglobin level | 2 years
  Change from baseline in hematological parameter
Measurement of absolute neutrophil count | 2 years
  Change from baseline in hematological parameter
Measurement of platelet count | 2 years
  Change from baseline in hematological parameter
IPMDS (International Pediatric Mitochondrial Disease Scale) | 2 years
  To compare the change in International Pediatric Mitochondrial Disease Scale (IPMDS) score during a follow up period of 3, 6 12 and 24 months post treatment. IPMDS total score ranges from 0 to 243. The score is expressed as the percentage of items which were feasible to perform. The lower the score is, the higher the child's function
Performance Score | 2 years
  Stabilization or improvement in performance score (Lansky score (for patients younger than 15 years) or Karnofsky (for patients older than 15) score relative to baseline
PEDI: Pediatric Evaluation of Disability Inventory | 2 years
  Stabilization or improvement in PEDI score relative to baseline
6-minute walk test | 2 years
  Stabilization or improvement in 6-minute walk test relative to baseline
30 Second chair stand | 2 years
  Stabilization or improvement in 30 Second chair stand relative to baseline
Hospitalization events | 1 year
  Reduction in number, cause and duration of hospitalization events relative to 12 months before IP treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center - Tel Ashomer, Ramat Gan, Israel